CLINICAL TRIAL: NCT06309537
Title: Chemoreflex Sensitivity in Heart Failure With Preserved Ejection Fraction
Brief Title: Chemoreflex Sensitivity in HFpEF
Acronym: CHEMO-HFpEF
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C830
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF: symptomatic patients with heart failure with preserved ejection fraction
  Interventions: Diagnostic Test: chemoreflex evaluation
- asymptomatic PH-LHD: asymptomatic left ventricular diastolic dysfunction with echocardiographic signs of pulmonary hypertension
  Interventions: Diagnostic Test: chemoreflex evaluation
- healthy volonteers
  Interventions: Diagnostic Test: chemoreflex evaluation

INTERVENTIONS:
Diagnostic Test: chemoreflex evaluation — the ventilatory response to carbon dioxide and hypoxia will be assessed in study participants

SUMMARY:
Patients with heart failure and a preserved left ventricular ejection fraction (HFpEF) almost invariably complain of exertional breathlessness. Abnormal cardiac hemodynamics with pulmonary congestion are believed to trigger dyspnea in this patients. However, some patients may complain of exertional breathlessness which seems to be out of proportion as compared with hemodynamic abnormalities.

Chemoreflex sensitivity accounts for the ventilatory responses to a variety of chemical stimuli, including carbon dioxide produced by the organism during exercise. Chemoreflex sensitivity can be augmented in heart failure with reduced left ventricular ejection fraction, and an increased chemoreflex sensitivity has been linked to symptoms, neurohumoral activation, breathing disturbances, and adverse prognosis.

However, the clinical correlates and implications of chemoreflex sensitivity in HFpEF have not been accurately studied.

We aim to characterize chemoreflex sensitivity in patients with a diagnosis of HFpEF, and to correlate chemoreflex sensitivity with clinical and hemodynamic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of symptomatic HFpEF (group 1)
* diagnosis of asymptomatic left ventricular diastolic dysfunction with echocardiographic signs of PH (group 2)
* healthy volunteers (group 3)

Exclusion Criteria:

* breastfeeding or childbearing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: we will include
  * symptomatic patients with a diagnosis of HFpEF
  * asymptomatic individuals with echocardiographic signs of PH attributable to left ventricular diastolic dysfynction
  * healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
difference in chemoreflex sensitivity between HFpEF and healthy controls | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Luca IRCCS Istituto Auxologico Italiano, Milan, Italy